CLINICAL TRIAL: NCT05146999
Title: A Phase 3b, Randomized, Double-Blind, Placebo-Controlled Study to Assess Aesthetic Improvement and Onset of QM1114-DP Treatment Effect in Subjects With Moderate to Severe Glabellar Lines
Brief Title: Assess Aesthetic Improvement and Onset of QM1114-DP in Subjects With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 43QM2106
Record Dates: First submitted 2021-10-31; First posted 2021-12-07 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Glabellar Frown Lines

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active arm - QM1114-DP (Active Comparator): a Botulinum Toxin Type A (BoNT-A)
  Interventions: Biological: QM1114-DP
- Inactive arm - Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: QM1114-DP — QM1114-DP
  Arms: Active arm - QM1114-DP
Biological: Placebo — Placebo
  Arms: Inactive arm - Placebo

SUMMARY:
The objective of this study is to evaluate the aesthetic improvement and onset of QM1114-DP treatment for subjects with moderate to severe glabellar lines

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years or older
* Moderate to severe GL at maximum frown as assessed by the Investigator
* Moderate to severe GL at maximum frown as assessed by the subject

Exclusion Criteria:

* Previous use of any botulinum toxin in facial areas within 9 months prior to study treatment
* Female who is pregnant, breast feeding or intends to conceive a child during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Galderma Research Site, Homewood, Alabama
  - Galderma Research Site, Manhattan Beach, California
  - Galderma Research Site, Vista, California
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, Hunt Valley, Maryland
  - Galderma Research Site, Omaha, Nebraska
  - Galderma Research Site, Chapel Hill, North Carolina
  - Galderma Research Site, Pflugerville, Texas
  - Galderma Research Site, Spring, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 9 investigational centers in the United States (US) from 09 May 2022 to 01 September 2023.
Pre-assignment Details: A total of 132 participants were enrolled and treated in this study.
Groups:
- Experimental: QM1114-DP: Participants received a single dose of 50 U (0.5 mL) (Milliliter) QM1114-DP intramuscularly (IM), divided into 5 equal aliquots injected into the glabellar area (10 U [0.1 mL] per injection point).
- Placebo Comparator: Placebo: Participants received a single dose of 0.5 mL placebo IM, divided into 5 equal aliquots injected into the glabellar area (0.1 mL per injection point).
Period: Overall Study
Arm/Group | Experimental: QM1114-DP | Placebo Comparator: Placebo
Started | 99 | 33
Completed | 89 | 27
Not Completed | 10 | 6
Not completed — Withdrew consent | 6 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants who were randomized and analyzed according to the treatment they were randomized based on the randomization scheme.
Groups:
- Experimental: QM1114-DP: Participants received a single dose of 50 U (0.5 mL) QM1114-DP IM, divided into 5 equal aliquots injected into the glabellar area (10 U [0.1 mL] per injection point).
- Total: Total of all reporting groups
Arm/Group | Experimental: QM1114-DP | Placebo Comparator: Placebo | Total
Number analyzed (Participants) | 99 | 33 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.72) | 52.5 (10.31) | 52.2 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 31 | 125
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 13 | 47
  Not Hispanic or Latino | 65 | 20 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 1 | 1
  White | 92 | 31 | 123
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders Using the Global Aesthetic Improvement Scale (GAIS) at Month 1
Description: Participant assessment at Month 1 of aesthetic change from baseline of the treated areas using the Global Aesthetic Improvement Scale. GAIS is a 7-graded scale: Very much worse; much worse; worse; no change; improved; much improved; or very much improved. A responder was defined as a participant who responded "improved," "much improved," or "very much improved" on the participant GAIS at maximum frown. Missing data is imputed as no change (non-responder).
Time Frame: At Month 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: QM1114-DP | Placebo Comparator: Placebo
Number analyzed (Participants) | 99 | 33
Participants | 92 | 3
Statistical Analysis 1: Comparison: Experimental: QM1114-DP vs Placebo Comparator: Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Treatment difference = 83.8, 95% CI 2-sided [72.81 to 94.87]

2. Secondary Outcome: Percentage of Participants Reporting Onset of Treatment Effect Using the Diary Card
Description: Following treatment at baseline, participants were asked to record their assessment of study treatment response in a diary card on Days 0 through 7. They were asked to respond "yes" or "no" to the following question: "Since being injected, have you noticed an improvement in the appearance of your glabellar lines (lines between your eyebrows) when you frown?" Response to treatment effect given by a Participant on first day as "yes" to the diary question.
Time Frame: At Days 0 through 7 post-treatment
Population: ITT population included all participants who were randomized and analyzed according to the treatment they were randomized based on the randomization scheme.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: QM1114-DP | Placebo Comparator: Placebo
Number analyzed (Participants) | 99 | 33
Participants | 89 | 3

3. Secondary Outcome: Number of Responders Using the Global Aesthetic Improvement Scale (GAIS) From Day 1 Through Month 12
Description: Participant assessment From Day 1 through Month 12 of aesthetic change from baseline of the treated areas using the Global Aesthetic Improvement Scale. GAIS is a 7-graded scale: Very much worse; much worse; worse; no change; improved; much improved; or very much improved. A responder was defined as a Participant who responded "improved," "much improved," or "very much improved" on the GAIS at maximum frown. This analysis is based on observed cases.
Time Frame: From Day 1 through Month 12
Population: ITT population included all participants who were randomized and analyzed according to the treatment they were randomized based on the randomization scheme. Here, "number analyzed" signifies participants in total observed cases at given time points.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Experimental: QM1114-DP | Placebo Comparator: Placebo
Number analyzed (Participants) | 99 | 33
participants
  Day 1: number analyzed (Participants) | 98 | 33
  Day 1 | 39 [30.10 to 49.49] | 4 [0.99 to 23.26]
  Day 2: number analyzed (Participants) | 98 | 32
  Day 2 | 66 [58.06 to 76.63] | 4 [1.04 to 23.96]
  Day 3: number analyzed (Participants) | 97 | 31
  Day 3 | 79 [73.71 to 89.18] | 4 [1.10 to 24.70]
  Day 4: number analyzed (Participants) | 96 | 31
  Day 4 | 87 [84.79 to 96.46] | 4 [1.10 to 24.70]
  Month 1: number analyzed (Participants) | 98 | 31
  Month 1 | 92 [89.13 to 98.62] | 3 [0.00 to 20.08]
  Month 3: number analyzed (Participants) | 98 | 30
  Month 3 | 87 [82.53 to 95.03] | 1 [0.00 to 9.76]
  Month 6: number analyzed (Participants) | 94 | 30
  Month 6 | 64 [58.66 to 77.51] | 1 [0.00 to 9.76]
  Month 7: number analyzed (Participants) | 91 | 29
  Month 7 | 51 [45.85 to 66.24] | 1 [0.00 to 10.09]
  Month 8: number analyzed (Participants) | 91 | 27
  Month 8 | 45 [39.18 to 59.72] | 1 [0.00 to 10.83]
  Month 9: number analyzed (Participants) | 89 | 27
  Month 9 | 38 [32.42 to 52.97] | 1 [0.00 to 10.83]
  Month 10: number analyzed (Participants) | 86 | 27
  Month 10 | 32 [26.99 to 47.43] | 0 [0.00 to 0.00]
  Month 11: number analyzed (Participants) | 86 | 26
  Month 11 | 31 [25.90 to 46.19] | 0 [0.00 to 0.00]
  Month 12: number analyzed (Participants) | 90 | 29
  Month 12 | 34 [27.76 to 47.79] | 1 [0.00 to 10.09]

ADVERSE EVENTS:
Time Frame: From Day 1 up to end of study (Up to 12 Months)
Description: Safety population included all participants who were treated with QM1114-DP and Placebo.
Arm/Group | Experimental: QM1114-DP | Placebo Comparator: Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/33
Other Adverse Events (participants affected / at risk) | 39/99 | 7/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: QM1114-DP (N=99) | Placebo Comparator: Placebo (N=33)
COVID-19 (Infections and infestations) | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Headache (Nervous system disorders) | 6 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Injection site bruising (General disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT05146999/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT05146999/SAP_001.pdf